CLINICAL TRIAL: NCT01326988
Title: Feasibility Study of the Use of Real-time Ultrasound Guidance to Administer Spinal Anesthesia
Brief Title: Real-time Ultrasound-guided Spinal Anesthesia:A Feasibility Study
Status: Completed | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Other Study IDs: Real-time Spinal Ultrasound
Record Dates: First submitted 2011-03-23; First posted 2011-03-31 (Estimated); Last update posted 2012-02-06 (Estimated); Status verified 2012-02

CONDITIONS: Ultrasound Spinal Anesthesia
Keywords: Spinal anesthesia; ultrasound; real-time

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients requiring spinal anesthesia for lower limb surgery: Patients of at least 18 years of age undergoing spinal anesthesia for elective lower limb surgery will be recruited. Therefore inclusion and exclusion criteria are the same as for traditionally administered spinal anesthesia as below. Additionally we will exclude those patients who are incapable of providing fully informed consent, patients who are currently enrolled in other studies and patients with communication difficulties
  Interventions: Procedure: Real-time ultrasound guided spinal anesthesia

INTERVENTIONS:
Procedure: Real-time ultrasound guided spinal anesthesia — The neuraxial US scan will be performed with the patient in the sitting or lateral position with the hip and knees slightly flexed using full aseptic technique. The spinal needle will be inserted in real-time under direct ultrasound guidance to administer the spinal anesthetic.

SUMMARY:
The traditional landmarks to locate the injection site and orientation of the spinal needle for spinal anesthesia are based on palpation of surface bony landmarks. However the actual injection target into the CSF is located at an unknown depth inside the patients 3 dimensional spinal anatomy which can itself vary in its orientation relative to these surface markers.Also bony surface markers may not be palpable in some patients or the patient may have altered spinal alignment. Thus an already blind procedure can become even more misguided involving multiple trial and error needle insertions. On the other hand ultrasound allows visualisation of deep target structures which are impalpable, it allows assessment of spinal alignment and thus directs the orientation of the seeking needle more accurately. Performing US in real-time during needle insertion gives continuous feedback about the correct needle approach path which should reduce the number of blind needle passes.

ELIGIBILITY:
Inclusion Criteria:

* Consenting patients of at least 18 years of age undergoing spinal anesthesia for elective lower limb surgery

Exclusion Criteria (are as for Spinal anesthesia generally)

* Patient refusal
* Sepsis or local infection at the site of injection
* Hypovolemia
* Coagulopathy (INR ≥1.5, Platelets < 75X 109 /L, anticoagulant therapy)
* Indeterminate neurologic disease
* Increased intracranial pressure
* Local anesthetic allergy
* Infection distinct from the site of injection
* Unknown duration of surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting for elective lower limb orthopaedic surgery to a specialist orthopaedic hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-04; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Number of ventral passes of the spinal needle into the patient | Assessed at time of spinal anesthetic injection (baseline)
Rate of successful performance of real-time ultrasound guided spinal needle insertion | Assessed at time of spinal anesthetic injection (baseline)

SECONDARY OUTCOMES:
Time for the procedure from first needle contact to the skin to injection of the medication into the spinal canal | Assessed at time of spinal anesthetic injection (baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Paul McHardy, MD FRCPC BA, Principal Investigator — Sunnybrook Health Sciences Center; Patrick H Conroy, MB FFARCSI, Principal Investigator — Sunnybrook Health Sciences Center; Luyet Cedric, MD, Principal Investigator — Sunnybrook Health Sciences Center; colin McCartney, FRCPC, Principal Investigator — Sunnybrook Health Sciences Center
Locations (1):
- Holland Orthopaedic & Arthritic Center, Toronto, Ontario, Canada

REFERENCES:
- [Background] Furness G, Reilly MP, Kuchi S. An evaluation of ultrasound imaging for identification of lumbar intervertebral level. Anaesthesia. 2002 Mar;57(3):277-80. doi: 10.1046/j.1365-2044.2002.2403_4.x. PMID 11892638
- [Background] Grau T, Leipold RW, Conradi R, Martin E, Motsch J. Ultrasound imaging facilitates localization of the epidural space during combined spinal and epidural anesthesia. Reg Anesth Pain Med. 2001 Jan-Feb;26(1):64-7. doi: 10.1053/rapm.2001.19633. No abstract available. PMID 11172514
- [Background] Karmakar MK, Li X, Ho AM, Kwok WH, Chui PT. Real-time ultrasound-guided paramedian epidural access: evaluation of a novel in-plane technique. Br J Anaesth. 2009 Jun;102(6):845-54. doi: 10.1093/bja/aep079. Epub 2009 Apr 27. PMID 19398454
- [Background] Tran D, Kamani AA, Al-Attas E, Lessoway VA, Massey S, Rohling RN. Single-operator real-time ultrasound-guidance to aim and insert a lumbar epidural needle. Can J Anaesth. 2010 Apr;57(4):313-21. doi: 10.1007/s12630-009-9252-1. PMID 20196236
- [Background] Chin KJ, Chan VW, Ramlogan R, Perlas A. Real-time ultrasound-guided spinal anesthesia in patients with a challenging spinal anatomy: two case reports. Acta Anaesthesiol Scand. 2010 Feb;54(2):252-5. doi: 10.1111/j.1399-6576.2009.02112.x. Epub 2009 Oct 15. PMID 19839951